CLINICAL TRIAL: NCT03771846
Title: Hepatic Arterial Infusion Chemotherapy of Irinotecan, Oxaliplatin, 5-Fluorouracil and Leucovorin Versus Systemic Chemotherapy of Gemcitabine and Oxaliplatin for Unresectable Intrahepatic Cholangiocarcinoma
Brief Title: HAIC Versus Systemic Chemotherapy for Unresectable ICC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S035
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: intrahepatic cholangiocarcinoma; systemic chemotherapy; hepatic artery infusion chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Irinotecan; Oxaliplatin; Fluorouracil; Leucovorin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepatic artery infusion chemotherapy (Experimental): Participants received hepatic artery infusion chemotherapy of irinotecan, oxaliplatin, 5-fluorouracil and leucovorin
  Interventions: Drug: irinotecan, oxaliplatin , fluorouracil, and leucovorin
- Systemic chemotherapy (Active Comparator): Participants received systemic chemotherapy of gemcitabine and oxaliplatin
  Interventions: Drug: gemcitabine and oxaliplatin

INTERVENTIONS:
Drug: irinotecan, oxaliplatin , fluorouracil, and leucovorin — administration of irinotecan, oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
  Arms: Hepatic artery infusion chemotherapy
Drug: gemcitabine and oxaliplatin — administration of gemcitabine and oxaliplatin via vein
  Arms: Systemic chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy (HAIC) of irinotecan, oxaliplatin, 5-fluorouracil and leucovorin compared systemic chemotherapy of gemcitabine and oxaliplatin in patients with unresectable intrahepatic cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of ICC
* Patients must have at least one tumor lesion that can be accurately measured according to mRECIST criteria.
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* Without distant metastasis, but intrahepatic lymph node metastasis is allowed
* The following laboratory parameters:

Platelet count ≥ 50,000/μL Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 6 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 months
  OS was defined as the duration from the date of randomization until the date of death from any cause. Participants who were lost to follow-up were censored at the last date the participant was known to be alive, and participants who remained alive were censored at the time of data cutoff.

SECONDARY OUTCOMES:
Progression free survival | 12 months
  PFS was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST), or date of death, whichever occurred first.
Time to progression | 12 months
  TTP was defined as the time from the date of randomization to the date of first documentation of disease progression based on modified Response Evaluation Criteria in Solid Tumors (mRECIST).
Number of adverse events. | 30 days
  Postoperative adverse events were graded based on CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Ming Shi, Guangzhou, Guangdong